CLINICAL TRIAL: NCT02620982
Title: Low-Intensity Extracorporeal Shock Wave Therapy for the Treatment of Vasculogenic Erectile Dysfunction
Brief Title: ARIES for Vasculogenic Erectile Dysfunction
Acronym: AriesIDE#1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dornier MedTech Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G140216
Record Dates: First submitted 2015-11-04; First posted 2015-12-03 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction, Physiological
Keywords: Shockwave; vascular ED; Organic ED
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARIES Application (Experimental): Low intensity Extracorporeal Shockwave Application utilizing the Dornier Aries
  Interventions: Device: ARIES (Extracorporal Shock Wave Application)

INTERVENTIONS:
Device: ARIES (Extracorporal Shock Wave Application) — The treatment protocol includes 1 treatment per week for 6 weeks and an application of 5000 shockwaves per session in 5 treatment areas with 1000 SW each at energy level 4-5 (energy flux density (0.051-0.062 mJ/mm²), while moving the applicator along the penile shaft within the treatment areas. The maximum energy applied during this treatment would be 23.35J.

SUMMARY:
This study aims to evaluate the safety and efficacy of low-intensity extracorporeal shock wave therapy utilizing the Dornier Aries in the treatment of erectile dysfunction of vasculogenic origin.

DETAILED DESCRIPTION:
An increasing number of men are suffering from the effects of Erectile Dysfunction (ED) each year. The development of oral therapies (phosphodiesterase 5 inhibitors) has been successful for many with the disease. However, these drugs may be contraindicated in patients with cardiovascular risk factors (which are often predecessors to developing ED) and are often ineffective in patients with other comorbid conditions, such as diabetes mellitus. The main objective of this study is to determine the safety and efficacy of low-intensity extracorporeal shock wave therapy using the Dornier Aries in the treatment of erectile dysfunction of vasculogenic origin.

This protocol allows for treatment of 23 men with 21-75 years of age with vasculogenic erectile dysfunction of at least 6 months' duration with low intensity extracorporeal shock wave therapy utilizing the Dornier Aries device.

This protocol includes the application of 5000 shockwaves per session in 5 treatment areas with 1000 SW each at energy level 4-5 (energy flux density (0.051-0.062 mJ/mm²), while moving the applicator along the penile shaft within the treatment areas. The maximum energy applied during this treatment would be 23.35J.

Conversely, the treatment protocol described within is designed to actually restore penile function as a disease-modifying therapy, and is not expected to require a maintenance regimen or continued treatments, as previous studies have demonstrated retained benefits at six months after the end of treatments.

Dornier MedTech hired an independent party to monitor data and perform internal audits to ensure the precision, quality, and integrity of the data collected. The investigator(s) agrees to permit access to study records, source data, and source documents for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 75 years
* Presence of Erectile Dysfunction for at least 6 months
* Having some response to a PDE5i or injection therapy (ICI) without penile scarring
* Vasculogenic ED
* IIEF-ED score ≥11 up to ≤25 while taking PDE5i or on ICI
* In a stable heterosexual relationship of more than three months' duration
* Agree to suspend all ED therapy for duration of study
* Agree to maintain their normal sexual habits
* Consent to participate

Exclusion Criteria:

* Radical prostatectomy
* Previous radiation therapy to pelvis
* Previous stem cell or platelet rich plasma therapy
* Previous pelvic surgeries
* Untreated Hypogonadism or thyroid disease
* Hormone usage, other than testosterone, clomiphene or thyroid medication
* Illicit drug usage as demonstrated in the drug screen
* Psychogenic ED
* Peyronie's Disease or penile curvature that negatively influences sexual activity
* Current anticoagulation therapy or significant hematological conditions

Ages: 21 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Changes in the mean of the International Index of Erectile Function ED Domain ("IIEF-ED") scores, in the absence of severe adverse events. | 1 month and 3 months
  Changes in the mean of the International Index of Erectile Function ED Domain ("IIEF-ED") scores, in the absence of severe adverse events. Higher scores indicate improved functionality according to the minimal clinically important difference (MCID) in erectile function from Rosen et al. 2011.

SECONDARY OUTCOMES:
Changes in penile base and tip rigidity | 3 months
  Changes in penile base and tip rigidity as measured by penile plethysmography (Rigiscan) of the penis will be evaluated and reported.
Changes in penile cavernosal artery peak systolic velocity (PSV) in [cm/s] by Penile doppler ultrasonography | 3 months
  Changes in penile cavernosal artery peak systolic velocity in [cm/s] as determined by color measurement of Penile doppler ultrasonography
Changes in penile corporal fibrosis | 1 month, 3 months
  changes in penile corporal fibrosis as determined by gray scale assessment as measured by duplex ultrasound of the penis during pharmacologic erection will be evaluated and reported
Changing in Erection Hardness score (EHS) | 1 month, 3 months
  EHS increase in patients with EHS < 2.
Changes in mean scores of the entire IIEF | 1 month, 3 months
  Changes in mean scores of the entire IIEF will be evaluated and reported.
Changes in mean scores of the SEP | 1 month, 3 months
  Changes in mean scores of Sexual Encounter Profile (SEP); [Unit on a Scale], will be evaluated and reported.
Changes in mean scores of the GAQ | 1 month, 3 months
  Changes in mean scores of Global Assessment Questionnaire (GAQ); [Unit on a Scale], common, will be evaluated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, M. D., Principal Investigator — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

REFERENCES:
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Vardi Y, Appel B, Kilchevsky A, Gruenwald I. Does low intensity extracorporeal shock wave therapy have a physiological effect on erectile function? Short-term results of a randomized, double-blind, sham controlled study. J Urol. 2012 May;187(5):1769-75. doi: 10.1016/j.juro.2011.12.117. Epub 2012 Mar 15. PMID 22425129
- [Background] Yee CH, Chan ES, Hou SS, Ng CF. Extracorporeal shockwave therapy in the treatment of erectile dysfunction: a prospective, randomized, double-blinded, placebo controlled study. Int J Urol. 2014 Oct;21(10):1041-5. doi: 10.1111/iju.12506. Epub 2014 Jun 17. PMID 24942563
- [Background] Assmus B, Walter DH, Seeger FH, Leistner DM, Steiner J, Ziegler I, Lutz A, Khaled W, Klotsche J, Tonn T, Dimmeler S, Zeiher AM. Effect of shock wave-facilitated intracoronary cell therapy on LVEF in patients with chronic heart failure: the CELLWAVE randomized clinical trial. JAMA. 2013 Apr 17;309(15):1622-31. doi: 10.1001/jama.2013.3527. PMID 23592107